CLINICAL TRIAL: NCT06412094
Title: A Comparative Controlled Study of the Effectiveness of Using a Mobile Application in Managing Pediatric Atopic Dermatitis
Brief Title: Use of a Mobile Health App in Managing Pediatric Atopic Dermatitis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Avanta Trading Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 242-SSMU
Record Dates: First submitted 2024-05-05; First posted 2024-05-14 (Actual); Last update posted 2024-05-14 (Actual); Status verified 2024-04

CONDITIONS: Atopic Dermatitis
MeSH Terms: conditions — Dermatitis, Atopic | interventions — Standard of Care

STUDY DESIGN:
Intervention Model Description: randomized controlled study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Standard care (Sham Comparator): Upon enrollment in the study at the end of the screening visit, participants in all groups receive a recommended treatment plan, according to the clinical severity of the AD, and. are instructed to contact the doctor via messenger for any questions related to their treatment.
  Interventions: Other: Standard care
- Standard care with access to the "AtopicApp" mobile application (Active Comparator): Subjects in the experimental and observational groups receive access to the "AtopicApp" mobile application, in addition to receiving standard medical care.
  Interventions: Other: Standard care; Behavioral: Access to the "AtopicApp" mobile application
- Standard care with access to the "AtopicApp" mobile application with potential virtual oversight (Experimental): The experimental group receives standard medical care, the AtopicApp mobile application, and information about doctor's virtual oversight through the app (monitoring registration and usage).
  Interventions: Other: Standard care; Behavioral: Access to the "AtopicApp" mobile application; Behavioral: Virtual oversight through the AtopicApp

INTERVENTIONS:
Other: Standard care — Recommendation of standard treatment plan, according to the clinical severity of the AD, and. are instruction to contact the doctor via messenger for any questions related to treatment recommendations.
Behavioral: Access to the "AtopicApp" mobile application — Access to the "AtopicApp" mobile application with 1 day after enrollment.
  Arms: Standard care with access to the "AtopicApp" mobile application; Standard care with access to the "AtopicApp" mobile application with potential virtual oversight
Behavioral: Virtual oversight through the AtopicApp — Notification of doctor's virtual oversight through the AtopicApp mobile application.
  Arms: Standard care with access to the "AtopicApp" mobile application with potential virtual oversight

SUMMARY:
A randomized controlled study in children with AD, divided into three groups: a control group without access to the app, an experimental observational group with the app, and an experimental interventional group with potential investigator supervision. Outcome measures included the SCORAD and the POEM scores.

DETAILED DESCRIPTION:
Three study groups: a control group that did not use the mobile health Atopic App, an experimental observational group provided with the mobile app without supervision by the investigators and experimental interventional group provided with the mobile app with potential supervision by the investigators. Upon study enrollment, participants receive recommended treatment plans and instructions for contacting the doctor via messenger for any questions during treatment. Virtual oversight disclosed to participant of the intervention arm, including registration status and regularity of use of the app.

Outcome endpoints are objective severity assessment using the SCORAD scale, and subjective assessment of effectiveness using the POEM scale.

ELIGIBILITY:
Inclusion Criteria:

* Children with AD and their parents that provided an informed consent to participate in the study

Exclusion Criteria:

* previous experience with the Atopic App
* participation in affiliated online Atopic School program
* presence of concomitant skin disease or pathological conditions that may affect the assessment of effectiveness (severe somatic diseases, mental disorders, oncologic or acute infectious diseases, etc.)
* avoidance from registration during consecutive 5 days following the screening visit (for participants in groups 2 or 3,)

Ages: 4 Months to 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 66 (Actual)
Dates: Start 2022-03-01 (Actual); Primary Completion 2022-12-26 (Actual); Study Completion 2022-12-26 (Actual)

PRIMARY OUTCOMES:
Patient Oriented Eczema Measure (POEM) | At baseline (screening visit, Day 1) and every 3 months thereafter (visits 1 and 2).
  A subjective tool that focuses on severity of atopic dermatitis as experienced by the patient. POEM scores can range from 0 to 28 (higher score reflects worse severity)
SCORAD (SCORing Atopic Dermatitis) | At baseline (screening visit, Day 1) and every 3 months thereafter (visits 1 and 2).
  A clinical tool for assessing the disease severity and subjective symptoms of atopic dermatitis. The SCORAD score range is between 0 and 103 points (higher score reflects worse severity).

CONTACTS AND LOCATIONS:
Overall Officials: Natalia Migacheva, MD, PhD, Principal Investigator — Samara State Medical University
Locations (1):
- Samara State Medical University, Samara, Russia

IPD SHARING:
Plan to Share IPD: Yes
De-identified IPD will be available to qualified researchers upon request by email to the principal investigator.
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: March 2024
Access Criteria: Upon request from an interested researcher